CLINICAL TRIAL: NCT01098006
Title: A Study in Adult Subjects With Chronic Hepatitis B Infection to Support the Development of Immunological Assays
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 113854
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Results first posted 2017-12-18 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Immunologic Tests
Keywords: Immunological assays; Chronic hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Immune tolerant patients Group (Other): Immune tolerant patients aged between and including 18 and 65 years of age at study start, having high levels of hepatitis B viruss (HBV) replication characterized by elevated HBV DNA levels and presence of hepatitis B envelope antigen (HBeAg), but normal alanine aminotransferase (ALT) levels with normal or mild histology findings.
  Interventions: Other: Blood withdrawal
- HBeAg positive Group (Other): HBeAg positive chronic Hepatitis B patients aged between and including 18 and 65 years of age at study start, having elevated or fluctuating ALT levels, presence of HBeAg and variable HBV DNA on a high level, histology mainly with activee inflammation and varying degrees of liver fibbrosis.
  Interventions: Other: Blood withdrawal
- Inactive carriers Group (Other): Inactive carriers aged between and including 18 and 65 years of age at study start, having normal ALT levels, undetectable or low levels of serum HBV DNA; absence of HBeAg and presence of anti-HBe antibodies, histology with little or no inflammation and varying degrees of liver fibrosis.
  Interventions: Other: Blood withdrawal
- HBeAg negative Group (Other): HBeAg negative chronic Hepatitis B patients aged between and including 18 and 65 years of age at study start, having absence of HBeAg, presence of anti-HBe, elevated ALT and HBV DNA levels, histology with significant inflammatory changes, liver fibrosis and cirrhosis.
  Interventions: Other: Blood withdrawal

INTERVENTIONS:
Other: Blood withdrawal — A single blood sample was to be taken from all subjects at the study visit. No study-related treatment was given to the study participants.

SUMMARY:
The purpose of this study is to develop and characterize immunological assays on blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the subject.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* A male or female between, and including, 18 and 65 years of age at study start.
* Evidence of chronic hepatitis B infection as per medical record.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject has practiced adequate contraception for 30 day prior to study start.

In addition to these general inclusion criteria, subjects should satisfy ALL specific criteria according to the specified group maximum 6 months prior to Visit 1 as per medical records:

Group A: Immune tolerant patients

* Viral load: > 2x107 IU/mL of HBV DNA
* HBeAg positive
* Normal levels of ALT according to lab range Group B: HBeAg positive chronic hepatitis B patients
* Viral load: > 2x104 IU/mL of HBV DNA
* HBeAg positive
* Increased levels of ALT and/or evidence of chronic hepatitis on liver biopsy Group C: Healthy carriers
* Viral load: not exceeding 2x103 IU/mL of HBV DNA
* HBeAg negative
* Normal levels of ALT measured at least twice, at least 3 months apart, during the last 6 months Group D: HBeAg negative chronic hepatitis B patients
* Viral load: > 2x103 IU/mL of HBV DNA
* HBeAg negative
* Increased levels of ALT and/or evidence of chronic hepatitis on liver biopsy

Exclusion Criteria:

* Any hepatitis B specific treatment prior to blood sampling at Visit 1.
* Any known clinically significant anaemia or any other condition within 7 days prior to study entry (Visit 1) as per medical records that would preclude the drawing of blood as described in the protocol.
* Receipt of live attenuated vaccines within 30 days preceding the blood sampling at Visit 1 and the administration of a pandemic influenza vaccine within 21 days preceding the blood sampling at Visit 1.
* Receipt of blood products within 120 days prior to study entry (Visit 1).
* Receipt of immunoglobulins within 120 days prior to study entry (Visit 1).
* Receipt of interferon within 120 days prior to study entry (Visit 1).
* Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding study start, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* History of immunosuppressive or immune-mediated disorders including autoimmune diseases, human immunodeficiency virus (HIV) infection and hepatitis C infection, based on medical history and physical examination (no laboratory testing required).
* Pregnant or lactating female.
* History of malignancy (unless there has been surgical excision followed by a sufficient observation period, of at least 5 years, to give a reasonable assurance of sustained cure and which, in the estimate of the investigator, is not likely to recur during the study period).
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs (including chloroquine) within six months prior to the blood sampling at Visit 1 (for corticosteroids, this will mean prednisone ≥10 milligram/day (10 mg/day), or equivalent). Inhaled and topical steroids are allowed.
* History of type I or type II diabetes mellitus including cases controlled with diet alone (a subject with past gestational diabetes is eligible).
* History of major congenital defect.
* Subjects with a history of, or current, alcohol or substance abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-04-29 (Actual); Primary Completion 2012-02-20 (Actual); Study Completion 2012-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Brussels, Belgium

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study period (i.e., from study initiation until study completion) was approximately 22 months (i.e., from April-2010 until February-2012). The duration of the study was one day for each subject.
Pre-assignment Details: All 99 subjects enrolled in the study were included in the analysis.
Groups:
- Immune Tolerant Patients Group: Immune tolerant patients aged between and including 18 and 65 years of age at study start, having high levels of hepatitis B virus (HBV) replication characterized by elevated HBV DNA levels and presence of hepatitis B envelope antigen (HBeAg), but normal alanine aminotransferase (ALT) levels with normal or mild histology findings.
- HBeAg Positive Group: HBeAg positive chronic Hepatitis B patients aged between and including 18 and 65 years of age at study start, having elevated or fluctuating ALT levels, presence of HBeAg and variable HBV DNA on a high level, histology mainly with active inflammation and varying degrees of liver fibrosis.
Period: Overall Study
Arm/Group | Immune Tolerant Patients Group | HBeAg Positive Group | Inactive Carriers Group | HBeAg Negative Group
Started | 7 | 11 | 60 | 21
Completed | 7 | 11 | 60 | 21
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immune Tolerant Patients Group | HBeAg Positive Group | Inactive Carriers Group | HBeAg Negative Group | Total
Number analyzed (Participants) | 7 | 11 | 60 | 21 | 99
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.4 (6.0) | 34.0 (14.2) | 36.9 (8.7) | 39.7 (15.1) | 36.43 (11.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 25 | 5 | 37
  Male | 4 | 7 | 35 | 16 | 62
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic Ancestry: African heritage/African American | 5 | 2 | 31 | 9 | 47
  Geographic Ancestry: Asian-Central/South Asian heritage | 0 | 2 | 1 | 0 | 3
  Geographic Ancestry: Asian-East Asian heritage | 1 | 2 | 2 | 0 | 5
  Geographic Ancestry: White-Arabic/North African heritage | 0 | 0 | 11 | 7 | 18
  Geographic Ancestry: White-Caucasian/European heritage | 0 | 5 | 15 | 4 | 24
  Geographic Ancestry: Other: Kazakstan | 1 | 0 | 0 | 0 | 1
  Geographic Ancestry: Other: Latino | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Cluster of Differentiation 4 (CD4) + Forkhead Box p3 (Foxp3) + Expressing CD45RA and/or Human Leucocyte Antigen DR Complex (HLA-DR) and/or Inducible T Cell Co-stimulator (ICOS) and/or PD1
Description: The frequency was assessed based on the following range of markers: CD4, CD45RA, ICOS, HLA-DR, PD-1 and anti-Foxp3.
Time Frame: At the time of the visit for each subject (i.e., Day 0)
Population: The analysis was performed on the According-to-protocol (ATP) cohort for immunogenicity, which included all subjects who met all eligibility criteria, with a blood sample available, who had satisfied all specific criteria according to their specific group and with data available for the markers analyzed within this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Treg cells/million cells
Arm/Group | Immune Tolerant Patients Group | HBeAg Positive Group | Inactive Carriers Group | HBeAg Negative Group
Number analyzed (Participants) | 4 | 10 | 56 | 19
Treg cells/million cells
  CD4+FOXP3+ | 5.025 [4.53 to 5.295] | 6.275 [5.07 to 6.51] | 4.185 [3.39 to 6.16] | 4.93 [4 to 6.16]
  CD4+FOXP3+CD45RA+: number analyzed (Participants) | 4 | 10 | 52 | 19
  CD4+FOXP3+CD45RA+ | 16.7 [8.53 to 28.9] | 16 [9.79 to 29.1] | 18 [14.4 to 29.25] | 16.2 [10.4 to 25.4]
  CD4+FOXP3+CD45RA+HLADR+ICOS+PD1-: number analyzed (Participants) | 4 | 10 | 46 | 18
  CD4+FOXP3+CD45RA+HLADR+ICOS+PD1- | 0.1299 [0.0785 to 1.769] | 0.0702 [0.0001 to 0.122] | 0.1755 [0.07 to 0.3] | 0.113 [0.0001 to 0.261]
  CD4+FOXP3+CD45RA+HLADR+ICOS-PD1+: number analyzed (Participants) | 4 | 10 | 46 | 18
  CD4+FOXP3+CD45RA+HLADR+ICOS-PD1+ | 0.1191 [0.0001 to 0.2565] | 0.119 [0.0747 to 0.134] | 0.0762 [0.03 to 0.189] | 0.0885 [0.0001 to 0.158]
  CD4+FOXP3+CD45RA+HLADR+ICOS-PD1-: number analyzed (Participants) | 4 | 10 | 46 | 18
  CD4+FOXP3+CD45RA+HLADR+ICOS-PD1- | 0.9705 [0.1534 to 1.95] | 0.2905 [0.21 to 0.528] | 0.51 [0.232 to 0.902] | 0.388 [0.09 to 0.567]
  CD4+FOXP3+CD45RA+HLADR-ICOS+PD1+: number analyzed (Participants) | 4 | 10 | 46 | 18
  CD4+FOXP3+CD45RA+HLADR-ICOS+PD1+ | 0.1836 [0.0001 to 0.4805] | 0.0637 [0.0001 to 0.112] | 0.106 [0.0339 to 0.227] | 0.092 [0.0675 to 0.3]
  CD4+FOXP3+CD45RA+HLADR-ICOS+PD1-: number analyzed (Participants) | 4 | 10 | 46 | 18
  CD4+FOXP3+CD45RA+HLADR-ICOS+PD1- | 0.3915 [0.1665 to 0.9885] | 0.356 [0.0747 to 0.725] | 0.74 [0.244 to 1.43] | 0.3185 [0.151 to 0.68]
  CD4+FOXP3+CD45RA+HLADR-ICOS-PD1+: number analyzed (Participants) | 4 | 10 | 46 | 18
  CD4+FOXP3+CD45RA+HLADR-ICOS-PD1+ | 0.0723 [0.0327 to 0.1541] | 0.1245 [0.0001 to 0.18] | 0.0972 [0.0001 to 0.182] | 0.138 [0.07 to 0.358]
  CD4+FOXP3+CD45RA+HLADR-ICOS-PD1-: number analyzed (Participants) | 4 | 10 | 52 | 19
  CD4+FOXP3+CD45RA+HLADR-ICOS-PD1- | 14.8 [7.605 to 23.3] | 14.2 [8.82 to 27.9] | 15.985 [12.7 to 24.85] | 14.6 [9.04 to 21.7]
  CD4+FOXP3+CD45RA-HLADR+ICOS+PD1+: number analyzed (Participants) | 4 | 10 | 50 | 19
  CD4+FOXP3+CD45RA-HLADR+ICOS+PD1+ | 0.629 [0.1209 to 1.27] | 2.48 [1.21 to 3.42] | 1.85 [0.937 to 2.93] | 2.03 [1.22 to 4.61]
  CD4+FOXP3+CD45RA-HLADR+ICOS+PD1-: number analyzed (Participants) | 4 | 10 | 52 | 19
  CD4+FOXP3+CD45RA-HLADR+ICOS+PD1- | 18.8 [7.58 to 27.7] | 13.35 [9.41 to 20.7] | 17.15 [11.15 to 24] | 14.86 [9.81 to 19.4]
  CD4+FOXP3+CD45RA-HLADR+ICOS-PD1+: number analyzed (Participants) | 4 | 10 | 47 | 19
  CD4+FOXP3+CD45RA-HLADR+ICOS-PD1+ | 0.5645 [0.0596 to 2.92] | 0.478 [0.234 to 1.57] | 0.651 [0.177 to 0.944] | 1.03 [0.49 to 2.64]
  CD4+FOXP3+CD45RA-HLADR+ICOS-PD1-: number analyzed (Participants) | 4 | 10 | 51 | 19
  CD4+FOXP3+CD45RA-HLADR+ICOS-PD1- | 18.7 [7.21 to 29.4] | 5.065 [3.31 to 10.4] | 7.16 [4.72 to 12.7] | 11.6 [4.37 to 23.04]
  CD4+FOXP3+CD45RA-HLADR-ICOS+PD1+: number analyzed (Participants) | 4 | 10 | 49 | 19
  CD4+FOXP3+CD45RA-HLADR-ICOS+PD1+ | 0.6269 [0.0815 to 1.82] | 1.285 [0.844 to 2.17] | 1.26 [0.8 to 2.14] | 1.96 [0.859 to 3.43]
  CD4+FOXP3+CD45RA-HLADR-ICOS+PD1-: number analyzed (Participants) | 4 | 10 | 52 | 19
  CD4+FOXP3+CD45RA-HLADR-ICOS+PD1- | 6.39 [3.48 to 8.345] | 9.66 [4.71 to 22.1] | 10.57 [5.955 to 16.035] | 9.79 [6.84 to 14.4]
  CD4+FOXP3+CD45RA-HLADR-ICOS-PD1+: number analyzed (Participants) | 4 | 10 | 50 | 19
  CD4+FOXP3+CD45RA-HLADR-ICOS-PD1+ | 0.7075 [0.2181 to 6.6895] | 2.07 [1.43 to 3.45] | 1.815 [0.51 to 2.88] | 3.28 [1.77 to 4.67]
  CD4+FOXP3+CD45RA-HLADR-ICOS-PD1-: number analyzed (Participants) | 4 | 10 | 52 | 19
  CD4+FOXP3+CD45RA-HLADR-ICOS-PD1- | 27.85 [21.35 to 44.5] | 36.8 [23.5 to 41.9] | 29.85 [24.065 to 38.4] | 33.2 [22.1 to 36.4]
  CD4+FOXP3+HLADR+: number analyzed (Participants) | 4 | 10 | 52 | 19
  CD4+FOXP3+HLADR+ | 45.4 [25.025 to 56] | 25.75 [20.5 to 35.5] | 31.65 [24.1 to 40] | 36.6 [19.5 to 47.94]
  CD4+FOXP3+ICOS+: number analyzed (Participants) | 4 | 10 | 52 | 19
  CD4+FOXP3+ICOS+ | 28 [16.35 to 38.1] | 41.1 [18 to 51.5] | 33.795 [21.6 to 48.5] | 35.3 [24.3 to 38.67]
  CD4+FOXP3+PD1+: number analyzed (Participants) | 4 | 10 | 52 | 19
  CD4+FOXP3+PD1+ | 5.505 [1.3975 to 13.225] | 8.465 [7.04 to 12] | 6.98 [3.57 to 10.45] | 9.61 [7.08 to 17.1]
  CD4+polypositives FOXP3+CD45RA+HLADR+ICOS+PD1: number analyzed (Participants) | 4 | 10 | 46 | 18
  CD4+polypositives FOXP3+CD45RA+HLADR+ICOS+PD1 | 0.1167 [0.0556 to 0.46] | 0.209 [0.0804 to 0.36] | 0.1645 [0.0894 to 0.25] | 0.1935 [0.0675 to 0.5]

2. Primary Outcome: Frequency of CD4+Foxp3- Expressing CD45RA and/or HLADR and/or ICOS and/or PD1
Description: The frequency was assessed based on the following range of markers: CD4, CD45RA, ICOS, HLA-DR, PD-1 and anti-Foxp3.
Time Frame: At the time of the visit for each subject (i.e., Day 0)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Treg cells/million cells
Arm/Group | Immune Tolerant Patients Group | HBeAg Positive Group | Inactive Carriers Group | HBeAg Negative Group
Number analyzed (Participants) | 4 | 10 | 56 | 19
Treg cells/million cells
  CD4+FOXP3- | 94.95 [94.7 to 95.45] | 93.75 [93.6 to 94.9] | 95.88 [93.8 to 96.61] | 95 [93.8 to 96]
  CD4+FOXP3-CD45RA+ | 38.7 [23.69 to 41.75] | 44.3 [36.6 to 57.7] | 33.9 [22.13 to 41.6] | 30.2 [16.47 to 41.07]
  CD4+FOXP3-CD45RA+HLADR+ICOS+PD1- | 0.0995 [0.046 to 0.2155] | 0.1103 [0.0519 to 0.167] | 0.0853 [0.0346 to 0.1865] | 0.0297 [0.004 to 0.115]
  CD4+FOXP3-CD45RA+HLADR+ICOS-PD1+ | 0.2825 [0.127 to 0.4995] | 0.1695 [0.123 to 0.369] | 0.267 [0.109 to 0.983] | 0.232 [0.147 to 0.857]
  CD4+FOXP3-CD45RA+HLADR+ICOS-PD1- | 1.53 [0.7938 to 1.68] | 1.52 [0.951 to 3.3] | 1.71 [0.406 to 2.805] | 1.07 [0.424 to 1.89]
  CD4+FOXP3-CD45RA+HLADR-ICOS+PD1+ | 0.0895 [0.0265 to 0.346] | 0.0928 [0.0569 to 0.141] | 0.0873 [0.0413 to 0.3565] | 0.0976 [0.0273 to 0.598]
  CD4+FOXP3-CD45RA+HLADR-ICOS+PD1- | 1.33 [0.6668 to 3.695] | 1.84 [0.48 to 3.52] | 0.973 [0.325 to 2.895] | 0.357 [0.0525 to 0.957]
  CD4+FOXP3-CD45RA+HLADR-ICOS-PD1+ | 0.174 [0.1254 to 0.3645] | 0.193 [0.0875 to 1.15] | 0.2585 [0.126 to 4.37] | 0.368 [0.0837 to 12.58]
  CD4+FOXP3-CD45RA+HLADR-ICOS-PD1- | 32.15 [18.68 to 38] | 36.95 [32 to 54.5] | 23.8 [10.64 to 31.75] | 14.96 [4.58 to 26.8]
  CD4+FOXP3-CD45RA-HLADR+ICOS+PD1+ | 1.37 [0.8255 to 1.935] | 0.995 [0.469 to 1.54] | 1.026 [0.3795 to 1.835] | 0.994 [0.549 to 1.96]
  CD4+FOXP3-CD45RA-HLADR+ICOS+PD1- | 1.515 [0.6425 to 2.11] | 0.727 [0.567 to 0.903] | 0.789 [0.352 to 1.51] | 0.522 [0.01 to 1.48]
  CD4+FOXP3-CD45RA-HLADR+ICOS-PD1+ | 1.065 [0.944 to 1.23] | 0.8265 [0.59 to 1.28] | 0.8765 [0.3965 to 2] | 1.34 [0.837 to 2.51]
  CD4+FOXP3-CD45RA-HLADR+ICOS-PD1- | 1.755 [1.2135 to 2.83] | 0.979 [0.571 to 1.52] | 1.32 [0.591 to 2.805] | 0.989 [0.07 to 4.27]
  CD4+FOXP3-CD45RA-HLADR-ICOS+PD1+ | 1.935 [1.34 to 5.78] | 2.28 [1.04 to 3.28] | 2.485 [1.17 to 7.05] | 3.02 [1.66 to 9.15]
  CD4+FOXP3-CD45RA-HLADR-ICOS+PD1- | 7.985 [4.65 to 13.555] | 8.835 [3.38 to 12] | 7.965 [4.25 to 14] | 5.95 [0.11 to 9.55]
  CD4+FOXP3-CD45RA-HLADR-ICOS-PD1+ | 8.21 [4.49 to 10.285] | 6.2 [3.88 to 11.8] | 7.385 [3.62 to 13.25] | 14.1 [7.07 to 24.5]
  CD4+FOXP3-CD45RA-HLADR-ICOS-PD1- | 35.6 [27.95 to 54.7] | 27.95 [23.4 to 40.8] | 34.8 [19.6 to 43.425] | 37.7 [16.8 to 52.6]
  CD4+FOXP3-HLADR+ | 7.845 [5.62 to 9.685] | 6.22 [4.4 to 7.11] | 8.66 [5.26 to 10.95] | 7.65 [5.92 to 11.9]
  CD4+FOXP3-ICOS+ | 14.6 [8.77 to 27.3] | 16.95 [11.1 to 18.5] | 21.03 [8.915 to 32.525] | 12.2 [8.85 to 21.34]
  CD4+FOXP3-PD1+ | 14.6 [10.565 to 18] | 9.895 [9.12 to 21] | 14.17 [8.025 to 40.88] | 20.3 [13.9 to 59.51]
  CD4+polypositives FOXP3-CD45RA+HLADR+ICOS+PD1 | 0.0998 [0.0562 to 0.1525] | 0.069 [0.0394 to 0.148] | 0.0689 [0.0377 to 0.2355] | 0.0431 [0.028 to 0.124]

3. Primary Outcome: Frequency of CD4+Foxp3+ Expressing CD45RA and/or Glucocorticoid-induced Tumor Necrosis Factor Receptor-related Protein (GITR) and/or Proliferation Marker Ki67
Description: The frequency was assessed based on the following range of markers: CD4, CD45RA, GITR, anti-Foxp3 and Ki67.
Time Frame: At the time of the visit for each subject (i.e., Day 0)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Treg cells/million cells
Arm/Group | Immune Tolerant Patients Group | HBeAg Positive Group | Inactive Carriers Group | HBeAg Negative Group
Number analyzed (Participants) | 4 | 11 | 55 | 20
Treg cells/million cells
  CD4+FOXP3+ | 5.335 [3.875 to 7.105] | 5.82 [5.62 to 6.8] | 4.68 [3.77 to 5.97] | 5.37 [4.18 to 6.24]
  CD4+FOXP3+CD45RA+: number analyzed (Participants) | 4 | 11 | 51 | 19
  CD4+FOXP3+CD45RA+ | 12.85 [11.2 to 22.2] | 14.8 [5.9 to 32.8] | 18.2 [13.6 to 27.34] | 16.5 [8.58 to 29.3]
  CD4+FOXP3+CD45RA+GITR+KI67-: number analyzed (Participants) | 4 | 11 | 47 | 19
  CD4+FOXP3+CD45RA+GITR+KI67- | 0.2955 [0.0861 to 1.1145] | 0.429 [0.211 to 0.571] | 0.49 [0.269 to 0.74] | 0.399 [0.288 to 0.599]
  CD4+FOXP3+CD45RA+GITR-KI67+: number analyzed (Participants) | 4 | 11 | 47 | 19
  CD4+FOXP3+CD45RA+GITR-KI67+ | 0.0985 [0.0663 to 0.218] | 0.2085 [0.12 to 0.564] | 0.234 [0.14 to 0.448] | 0.267 [0.07 to 0.452]
  CD4+FOXP3+CD45RA+GITR-KI67-: number analyzed (Participants) | 4 | 11 | 51 | 19
  CD4+FOXP3+CD45RA+GITR-KI67- | 12.55 [10.75 to 20.55] | 13.8 [3.9 to 29.9] | 17.7 [13.1 to 25.7] | 15.4 [7.34 to 27.93]
  CD4+FOXP3+CD45RA-GITR+KI67+: number analyzed (Participants) | 4 | 11 | 51 | 19
  CD4+FOXP3+CD45RA-GITR+KI67+ | 9.26 [7.055 to 11.05] | 8.24 [4.47 to 10.4] | 8.14 [6.32 to 11.32] | 7.43 [5.09 to 9.56]
  CD4+FOXP3+CD45RA-GITR+KI67-: number analyzed (Participants) | 4 | 11 | 51 | 19
  CD4+FOXP3+CD45RA-GITR+KI67- | 35.65 [26.5 to 43.5] | 33.4 [21.6 to 45.2] | 27.34 [22.3 to 34.18] | 28.8 [20 to 36.63]
  CD4+FOXP3+CD45RA-GITR-KI67+: number analyzed (Participants) | 4 | 11 | 51 | 19
  CD4+FOXP3+CD45RA-GITR-KI67+ | 4.84 [3.44 to 7.11] | 3.66 [2.58 to 5.58] | 4.69 [3.88 to 6.77] | 4.27 [3.67 to 6.19]
  CD4+FOXP3+CD45RA-GITR-KI67-: number analyzed (Participants) | 4 | 11 | 51 | 19
  CD4+FOXP3+CD45RA-GITR-KI67- | 30.9 [22.6 to 45.3] | 32.3 [24.4 to 36.7] | 37.1 [28.1 to 42.6] | 41.4 [36 to 47]
  CD4+FOXP3+GITR+: number analyzed (Participants) | 4 | 11 | 51 | 19
  CD4+FOXP3+GITR+ | 46.4 [34.95 to 55] | 49.1 [26.5 to 57.4] | 38.5 [30.51 to 46] | 36.9 [25.6 to 45.6]
  CD4+FOXP3+KI67+: number analyzed (Participants) | 4 | 11 | 51 | 19
  CD4+FOXP3+KI67+ | 13.95 [12.25 to 17.25] | 14.2 [8.14 to 15.7] | 13.8 [10.89 to 18.9] | 12.7 [9.49 to 16.5]
  CD4+polypositives FOXP3+CD45RA+GITR+KI67: number analyzed (Participants) | 4 | 10 | 47 | 19
  CD4+polypositives FOXP3+CD45RA+GITR+KI67 | 0.2685 [0.1568 to 0.4415] | 0.1855 [0.0945 to 0.42] | 0.331 [0.14 to 0.53] | 0.28 [0.175 to 0.512]

4. Primary Outcome: Frequency of CD4+Foxp3- Expressing CD45RA and/or GITR and/or Ki67
Description: The frequency was assessed based on the following range of markers: CD4, CD45RA, GITR, anti-Foxp3 and Ki67.
Time Frame: At the time of the visit for each subject (i.e., Day 0)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Treg cells/million cells
Arm/Group | Immune Tolerant Patients Group | HBeAg Positive Group | Inactive Carriers Group | HBeAg Negative Group
Number analyzed (Participants) | 4 | 11 | 55 | 20
Treg cells/million cells
  CD4+FOXP3- | 94.65 [92.85 to 96.15] | 94.2 [93.3 to 94.4] | 95.31 [94 to 96.2] | 94.65 [93.75 to 95.85]
  CD4+FOXP3-CD45RA+ | 45.95 [42.8 to 49.25] | 42.9 [29.4 to 56.5] | 34.3 [26.7 to 44.3] | 33.4 [24.295 to 43.4]
  CD4+FOXP3-CD45RA+GITR+KI67- | 0.6515 [0.4665 to 5.7485] | 0.567 [0.359 to 0.891] | 0.609 [0.27 to 2.23] | 0.563 [0.3155 to 1.46]
  CD4+FOXP3-CD45RA+GITR-KI67+ | 0.328 [0.226 to 0.393] | 0.365 [0.332 to 0.685] | 0.251 [0.142 to 0.404] | 0.2275 [0.166 to 0.471]
  CD4+FOXP3-CD45RA+GITR-KI67- | 42.85 [36.6 to 48.25] | 42.5 [27.8 to 55.2] | 30.14 [14.15 to 41.1] | 30.3 [19.95 to 37.9]
  CD4+FOXP3-CD45RA-GITR+KI67+ | 1.0535 [0.583 to 1.38] | 0.566 [0.472 to 0.974] | 0.854 [0.528 to 1.46] | 0.7955 [0.5645 to 1.27]
  CD4+FOXP3-CD45RA-GITR+KI67- | 13.35 [8.36 to 19.25] | 12.6 [4.34 to 15.6] | 12.94 [7.33 to 16.51] | 13.225 [9.03 to 14.95]
  CD4+FOXP3-CD45RA-GITR-KI67+ | 1.575 [1.405 to 2.05] | 1.56 [1.25 to 2.44] | 1.83 [1.29 to 2.24] | 1.455 [1.053 to 2.175]
  CD4+FOXP3-CD45RA-GITR-KI67- | 37.5 [29.1 to 45.8] | 43.7 [34.3 to 52.6] | 49.1 [40.7 to 58.5] | 50.9 [38.55 to 59.655]
  CD4+FOXP3-GITR+ | 15.05 [9.585 to 26.7] | 14 [5.88 to 17.1] | 15.9 [8.49 to 19.72] | 15.7 [10.155 to 17.65]
  CD4+FOXP3-KI67+ | 3.18 [2.47 to 3.98] | 3.42 [2.32 to 4] | 3.32 [2.43 to 4.57] | 3.28 [2.06 to 3.76]
  CD4+polypositives FOXP3-CD45RA+GITR+KI67 | 0.1275 [0.0874 to 0.331] | 0.0944 [0.081 to 0.162] | 0.0945 [0.049 to 0.202] | 0.0901 [0.0717 to 0.14]

5. Primary Outcome: Frequency of CD4+Foxp3+ Expressing CD45RA and/or, Chemokine (C-C Motif) Receptor 7 (CCR7) and/or CD62L
Description: The frequency was assessed based on the following range of markers: CD4, CD45RA, CCR7, CD62L and anti-Foxp3.
Time Frame: At the time of the visit for each subject (i.e., Day 0)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Treg cells/million cells
Arm/Group | Immune Tolerant Patients Group | HBeAg Positive Group | Inactive Carriers Group | HBeAg Negative Group
Number analyzed (Participants) | 4 | 11 | 57 | 19
Treg cells/million cells
  CD4+FOXP3+ | 4.12 [3.33 to 5.14] | 5.48 [4.56 to 6.07] | 4.26 [3.19 to 6] | 4.64 [2.87 to 5.22]
  CD4+FOXP3+CCR7+: number analyzed (Participants) | 4 | 11 | 48 | 18
  CD4+FOXP3+CCR7+ | 44.15 [38.45 to 50.9] | 48.4 [35.1 to 61.1] | 54.065 [43.54 to 59.75] | 42.4 [29.9 to 55.9]
  CD4+FOXP3+CCR7+CD45RA+CD62L-: number analyzed (Participants) | 4 | 10 | 46 | 18
  CD4+FOXP3+CCR7+CD45RA+CD62L- | 0.4295 [0.1971 to 0.515] | 0.2005 [0.0747 to 0.366] | 0.11 [0.0485 to 0.307] | 0.105 [0.0676 to 0.364]
  CD4+FOXP3+CCR7+CD45RA-CD62L+: number analyzed (Participants) | 4 | 11 | 48 | 18
  CD4+FOXP3+CCR7+CD45RA-CD62L+ | 27.85 [21.45 to 33.35] | 30.1 [22.6 to 32.6] | 34.66 [27.24 to 39.24] | 25.65 [21.4 to 31.7]
  CD4+FOXP3+CCR7+CD45RA-CD62L-: number analyzed (Participants) | 4 | 10 | 46 | 18
  CD4+FOXP3+CCR7+CD45RA-CD62L- | 1.73 [1.027 to 3.11] | 3.4 [1.56 to 4.86] | 1.88 [1.18 to 2.83] | 2.065 [1.63 to 2.76]
  CD4+FOXP3+CCR7-CD45RA+CD62L+: number analyzed (Participants) | 4 | 11 | 47 | 18
  CD4+FOXP3+CCR7-CD45RA+CD62L+ | 0.909 [0.2809 to 2.32] | 0.522 [0.224 to 2.14] | 0.59 [0.315 to 1.13] | 0.8925 [0.36 to 1.94]
  CD4+FOXP3+CCR7-CD45RA+CD62L-: number analyzed (Participants) | 4 | 10 | 46 | 18
  CD4+FOXP3+CCR7-CD45RA+CD62L- | 0.0502 [0.022 to 0.0671] | 0.0732 [0.0249 to 0.142] | 0.0499 [0.0001 to 0.0805] | 0.075 [0.0277 to 0.14]
  CD4+FOXP3+CCR7-CD45RA-CD62L+: number analyzed (Participants) | 4 | 11 | 48 | 18
  CD4+FOXP3+CCR7-CD45RA-CD62L+ | 43.3 [34.85 to 51.85] | 36.6 [31.7 to 43.5] | 37.7 [32.9 to 44.35] | 42.5 [32.6 to 56.08]
  CD4+FOXP3+CCR7-CD45RA-CD62L-: number analyzed (Participants) | 4 | 11 | 48 | 18
  CD4+FOXP3+CCR7-CD45RA-CD62L- | 9.6 [7.19 to 13.9] | 13.2 [6.19 to 16.8] | 6.56 [4.805 to 10.06] | 8.985 [6.93 to 15.9]
  CD4+FOXP3+CD45RA+: number analyzed (Participants) | 4 | 11 | 48 | 18
  CD4+FOXP3+CD45RA+ | 14.8 [13.5 to 19.65] | 14 [8.64 to 31.2] | 16.95 [11.8 to 23] | 14.25 [8.43 to 19.48]
  CD4+FOXP3+CD62L+: number analyzed (Participants) | 4 | 11 | 48 | 18
  CD4+FOXP3+CD62L+ | 88.55 [82.7 to 91.05] | 81.5 [77.7 to 92.2] | 90.85 [87.005 to 93.45] | 88.2 [78.3 to 91.2]
  CD4+polypositives FOXP3+CCR7+CD45RA+CD62L: number analyzed (Participants) | 4 | 11 | 48 | 18
  CD4+polypositives FOXP3+CCR7+CD45RA+CD62L | 14.25 [11.295 to 18.4] | 11.3 [5.76 to 28.6] | 15.1 [11.25 to 21.4] | 11.95 [6.42 to 15.28]

6. Primary Outcome: Frequency of CD4+Foxp3- Expressing CD45RA and/or CCR7 and/or CD62L
Description: The frequency was assessed based on the following range of markers: CD4, CD45RA, CCR7, CD62L and anti-Foxp3.
Time Frame: At the time of the visit for each subject (i.e., Day 0)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Treg cells/million cells
Arm/Group | Immune Tolerant Patients Group | HBeAg Positive Group | Inactive Carriers Group | HBeAg Negative Group
Number analyzed (Participants) | 4 | 11 | 57 | 19
Treg cells/million cells
  CD4+FOXP3- | 95.9 [94.85 to 96.7] | 94.4 [93.9 to 95.4] | 95.73 [94 to 96.8] | 95.4 [94.8 to 97.1]
  CD4+FOXP3-CCR7+ | 83.2 [75.3 to 84.1] | 79.5 [69.4 to 91.6] | 76.1 [67.8 to 83.2] | 70.8 [56.8 to 82.1]
  CD4+FOXP3-CCR7+CD45RA+CD62L- | 0.4295 [0.1966 to 0.6885] | 0.474 [0.259 to 0.664] | 0.305 [0.187 to 0.58] | 0.272 [0.196 to 1.03]
  CD4+FOXP3-CCR7+CD45RA-CD62L+ | 32.2 [25.45 to 38.3] | 26.7 [24.5 to 31.7] | 34.7 [26.7 to 40.32] | 33.4 [22.7 to 36.04]
  CD4+FOXP3-CCR7+CD45RA-CD62L- | 5.79 [3.915 to 7.415] | 4.09 [2.86 to 5.84] | 4.35 [2.5 to 6.33] | 5.16 [2.4 to 8.58]
  CD4+FOXP3-CCR7-CD45RA+CD62L+ | 1.005 [0.388 to 1.485] | 0.755 [0.259 to 2.1] | 0.719 [0.469 to 2.36] | 1.01 [0.415 to 2.12]
  CD4+FOXP3-CCR7-CD45RA+CD62L- | 1.2035 [0.594 to 2.06] | 1.72 [0.688 to 2.08] | 0.82 [0.466 to 1.88] | 0.855 [0.34 to 1.22]
  CD4+FOXP3-CCR7-CD45RA-CD62L+ | 7.91 [7.115 to 11.19] | 6.69 [3.54 to 9.01] | 8.86 [7.11 to 12.22] | 10.84 [5.57 to 16]
  CD4+FOXP3-CCR7-CD45RA-CD62L- | 7.795 [6.36 to 11.38] | 9.79 [5.37 to 14.7] | 10.54 [7.72 to 15.7] | 15.5 [6.36 to 18.6]
  CD4+FOXP3-CD45RA+ | 47.45 [39.4 to 49.5] | 47.2 [40.3 to 49.7] | 38.6 [30.79 to 48.05] | 33.8 [28.3 to 46.92]
  CD4+FOXP3-CD62L+ | 83.6 [81.4 to 85.95] | 85 [77.1 to 88.7] | 83.6 [76.4 to 86.3] | 75.3 [72 to 86]
  CD4+polypositives FOXP3-CCR7+CD45RA+CD62L | 44.45 [37.85 to 45.65] | 39.7 [23.4 to 48.2] | 35.56 [26.4 to 43.2] | 32.1 [21.6 to 41.29]

7. Primary Outcome: Frequency of CD4+Foxp3+ Expressing CD45RA and/or CD39 and/or Tumor Necrosis Factor Receptor 2 (TNFR2)
Description: The frequency was assessed based on the following range of markers: CD4, CD45RA, CD39, TNFR2 and anti-Foxp3.
Time Frame: At the time of the visit for each subject (i.e., Day 0)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Treg cells/million cells
Arm/Group | Immune Tolerant Patients Group | HBeAg Positive Group | Inactive Carriers Group | HBeAg Negative Group
Number analyzed (Participants) | 4 | 11 | 56 | 19
Treg cells/million cells
  CD4+FOXP3+ | 5.375 [3.745 to 6.185] | 5.68 [4.84 to 6.32] | 4.415 [3.195 to 5.995] | 5.32 [3.98 to 6.85]
  CD4+FOXP3+CD39+: number analyzed (Participants) | 4 | 11 | 50 | 19
  CD4+FOXP3+CD39+ | 47.25 [28.4 to 52.3] | 54.7 [24.1 to 65.5] | 42.2 [15.2 to 54.8] | 46.9 [32.9 to 63.79]
  CD4+FOXP3+CD39+CD45RA+TNFR2-: number analyzed (Participants) | 4 | 10 | 48 | 18
  CD4+FOXP3+CD39+CD45RA+TNFR2- | 0.0001 [0.0001 to 0.0161] | 0.0156 [0.0001 to 0.112] | 0.0381 [0.0001 to 0.0706] | 0.0001 [0.0001 to 0.0512]
  CD4+FOXP3+CD39+CD45RA-TNFR2+: number analyzed (Participants) | 4 | 11 | 50 | 19
  CD4+FOXP3+CD39+CD45RA-TNFR2+ | 45.55 [27.75 to 49.65] | 37.3 [23.6 to 63.8] | 39.85 [14.8 to 50.49] | 43.3 [31.3 to 61.6]
  CD4+FOXP3+CD39+CD45RA-TNFR2-: number analyzed (Participants) | 4 | 10 | 48 | 19
  CD4+FOXP3+CD39+CD45RA-TNFR2- | 0.48 [0.133 to 0.831] | 0.165 [0.12 to 0.352] | 0.1915 [0.0977 to 0.6025] | 0.32 [0.155 to 0.502]
  CD4+FOXP3+CD39-CD45RA+TNFR2+: number analyzed (Participants) | 4 | 11 | 50 | 19
  CD4+FOXP3+CD39-CD45RA+TNFR2+ | 14.8 [11.47 to 17.45] | 11 [8.25 to 24.8] | 17.075 [12.6 to 21.3] | 13.12 [6.96 to 18]
  CD4+FOXP3+CD39-CD45RA+TNFR2-: number analyzed (Participants) | 4 | 10 | 49 | 19
  CD4+FOXP3+CD39-CD45RA+TNFR2- | 1.009 [0.5365 to 1.325] | 0.7245 [0.497 to 1.16] | 0.815 [0.48 to 1.79] | 0.658 [0.155 to 1.81]
  CD4+FOXP3+CD39-CD45RA-TNFR2+: number analyzed (Participants) | 4 | 11 | 50 | 19
  CD4+FOXP3+CD39-CD45RA-TNFR2+ | 35.25 [30.15 to 56.35] | 25.4 [21.9 to 45.3] | 37.685 [28.4 to 56.7] | 32.01 [24.4 to 49]
  CD4+FOXP3+CD39-CD45RA-TNFR2-: number analyzed (Participants) | 4 | 10 | 50 | 19
  CD4+FOXP3+CD39-CD45RA-TNFR2- | 0.8705 [0.7215 to 1.256] | 0.6765 [0.448 to 0.776] | 1.085 [0.628 to 2.16] | 0.702 [0.4 to 1.84]
  CD4+FOXP3+CD45RA+: number analyzed (Participants) | 4 | 11 | 50 | 19
  CD4+FOXP3+CD45RA+ | 17 [13.1 to 20.05] | 13.4 [9.32 to 39.3] | 19.75 [15.8 to 24.5] | 15.7 [8.08 to 21.6]
  CD4+FOXP3+TNFR2+: number analyzed (Participants) | 4 | 11 | 50 | 19
  CD4+FOXP3+TNFR2+ | 97.7 [97.15 to 98] | 98.4 [98 to 98.6] | 97.25 [95.7 to 98.6] | 97.9 [96.2 to 98.9]
  CD4+pol FOXP3+CD39+CD45RA+TNFR2: number analyzed (Participants) | 4 | 10 | 48 | 18
  CD4+pol FOXP3+CD39+CD45RA+TNFR2 | 1.2415 [0.509 to 1.805] | 1.49 [1.09 to 2.25] | 1.215 [0.47 to 2.03] | 0.9295 [0.593 to 1.35]

8. Primary Outcome: Frequency of CD4+Foxp3- Expressing CD45RA and/or CD39 and/or TNFR2
Description: The frequency was assessed based on the following range of markers: CD4, CD45RA, CD39, TNFR2 and anti-Foxp3.
Time Frame: At the time of the visit for each subject (i.e., Day 0)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Treg cells/million cells
Arm/Group | Immune Tolerant Patients Group | HBeAg Positive Group | Inactive Carriers Group | HBeAg Negative Group
Number analyzed (Participants) | 4 | 11 | 56 | 19
Treg cells/million cells
  CD4+FOXP3- | 94.65 [93.8 to 96.3] | 94.3 [93.7 to 95.2] | 95.585 [94 to 96.8] | 94.7 [93.2 to 96]
  CD4+FOXP3-CD39+ | 3.395 [2.82 to 4.625] | 3.93 [1.55 to 5.16] | 4.015 [2.135 to 5.34] | 4.83 [3.7 to 6.05]
  CD4+FOXP3-CD39+CD45RA+TNFR2- | 0.828 [0.4515 to 1.41] | 0.531 [0.401 to 0.698] | 0.5295 [0.352 to 0.786] | 0.46 [0.31 to 0.64]
  CD4+FOXP3-CD39+CD45RA-TNFR2+ | 1.965 [0.936 to 2.65] | 2.25 [0.637 to 2.91] | 2.22 [0.7095 to 2.9] | 3.24 [1.85 to 4.15]
  CD4+FOXP3-CD39+CD45RA-TNFR2- | 0.6185 [0.3685 to 0.857] | 0.754 [0.133 to 0.898] | 0.6635 [0.2125 to 1.085] | 0.749 [0.547 to 1.04]
  CD4+FOXP3-CD39-CD45RA+TNFR2+ | 2.66 [1.79 to 4.095] | 2.55 [1.7 to 3.2] | 3.585 [2.115 to 4.485] | 3.04 [1.41 to 3.77]
  CD4+FOXP3-CD39-CD45RA+TNFR2- | 41.85 [36.5 to 45.7] | 40.9 [28.4 to 52.9] | 36.41 [29.9 to 47.9] | 29.9 [24.3 to 40.7]
  CD4+FOXP3-CD39-CD45RA-TNFR2+ | 30.2 [29.3 to 30.55] | 29.6 [19.6 to 36.3] | 32.155 [24.21 to 41.345] | 38.9 [26.2 to 46.1]
  CD4+FOXP3-CD39-CD45RA-TNFR2- | 22.9 [18.1 to 26.5] | 20 [16.4 to 23.1] | 21.42 [18.6 to 25.3] | 20.9 [17.95 to 25.6]
  CD4+FOXP3-CD45RA+ | 45.2 [40.15 to 50.6] | 48 [39.8 to 55.3] | 41.235 [33.795 to 52.195] | 33.8 [25.6 to 47.44]
  CD4+FOXP3-TNFR2+ | 35.05 [33.7 to 36.4] | 34.1 [24 to 50.2] | 39.23 [29.55 to 46.935] | 45.6 [33 to 53.2]
  CD4+polypositives FOXP3-CD39+CD45RA+TNFR2 | 0.3485 [0.209 to 0.561] | 0.252 [0.173 to 0.398] | 0.2795 [0.221 to 0.472] | 0.336 [0.244 to 0.478]

9. Primary Outcome: Frequency of CD4+Foxp3+ Expressing CD45RA and/or CTLA4 and/or OX40
Description: The frequency was assessed based on the following range of markers: CD4, CD45RA, CTLA4, OX40 and anti-Foxp3.
Time Frame: At the time of the visit for each subject (i.e., Day 0)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Treg cells/million cells
Arm/Group | Immune Tolerant Patients Group | HBeAg Positive Group | Inactive Carriers Group | HBeAg Negative Group
Number analyzed (Participants) | 4 | 11 | 56 | 18
Treg cells/million cells
  CD4+FOXP3+ | 5.555 [1.8151 to 8.095] | 6.09 [5.17 to 6.73] | 4.655 [3.38 to 6.145] | 5.045 [3.23 to 5.98]
  CD4+FOXP3+CD45RA+: number analyzed (Participants) | 3 | 11 | 51 | 17
  CD4+FOXP3+CD45RA+ | 17.8 [15.8 to 19.7] | 17.4 [7.16 to 22.8] | 18.5 [13.01 to 26.3] | 16.6 [8.81 to 24.5]
  CD4+FOXP3+CD45RA+CTLA4+OX40-: number analyzed (Participants) | 3 | 9 | 50 | 17
  CD4+FOXP3+CD45RA+CTLA4+OX40- | 1.5 [1.25 to 1.66] | 1.75 [1.24 to 2.63] | 1.32 [0.47 to 2.35] | 1.09 [0.74 to 2.4]
  CD4+FOXP3+CD45RA+CTLA4-OX40+: number analyzed (Participants) | 3 | 9 | 49 | 17
  CD4+FOXP3+CD45RA+CTLA4-OX40+ | 0.107 [0.0722 to 0.26] | 0.174 [0.106 to 0.205] | 0.11 [0.06 to 0.31] | 0.126 [0.06 to 0.252]
  CD4+FOXP3+CD45RA+CTLA4-OX40-: number analyzed (Participants) | 3 | 11 | 51 | 17
  CD4+FOXP3+CD45RA+CTLA4-OX40- | 15.9 [14 to 17.9] | 15.2 [5.85 to 20.9] | 16.1 [11.3 to 23.72] | 13.2 [6.32 to 21.9]
  CD4+FOXP3+CD45RA-CTLA4+OX40+: number analyzed (Participants) | 3 | 11 | 50 | 17
  CD4+FOXP3+CD45RA-CTLA4+OX40+ | 1.73 [1.3 to 2.53] | 2.08 [1.22 to 4.04] | 1.345 [0.631 to 2.13] | 2.38 [0.84 to 4.15]
  CD4+FOXP3+CD45RA-CTLA4+OX40-: number analyzed (Participants) | 3 | 11 | 51 | 17
  CD4+FOXP3+CD45RA-CTLA4+OX40- | 28.4 [25 to 30.4] | 41 [26.5 to 47.4] | 24.5 [15.9 to 38.3] | 31.7 [28.08 to 39.1]
  CD4+FOXP3+CD45RA-CTLA4-OX40+: number analyzed (Participants) | 3 | 10 | 50 | 17
  CD4+FOXP3+CD45RA-CTLA4-OX40+ | 8.16 [6.28 to 11.9] | 1.915 [0.872 to 3.26] | 1.515 [0.62 to 2.54] | 1.39 [0.586 to 1.98]
  CD4+FOXP3+CD45RA-CTLA4-OX40-: number analyzed (Participants) | 3 | 11 | 51 | 17
  CD4+FOXP3+CD45RA-CTLA4-OX40- | 43.9 [39.5 to 47.5] | 42 [26.4 to 47.3] | 47.9 [39.5 to 56.2] | 38.1 [32.6 to 49.3]
  CD4+FOXP3+CTLA4+: number analyzed (Participants) | 3 | 11 | 51 | 17
  CD4+FOXP3+CTLA4+ | 31.8 [27.9 to 34.6] | 45 [31.8 to 53.5] | 27.5 [17.64 to 40.9] | 39.3 [32.1 to 51.2]
  CD4+FOXP3+OX40+: number analyzed (Participants) | 3 | 11 | 51 | 17
  CD4+FOXP3+OX40+ | 10.1 [8.15 to 14.7] | 5.15 [2.68 to 6.51] | 3.66 [1.72 to 6.15] | 3.94 [2.16 to 7.55]
  CD4+polypositives FOXP3+CD45RA+CTLA4+OX40: number analyzed (Participants) | 3 | 10 | 50 | 17
  CD4+polypositives FOXP3+CD45RA+CTLA4+OX40 | 0.188 [0.0722 to 0.364] | 0.118 [0.0709 to 0.381] | 0.19 [0.0322 to 0.37] | 0.283 [0.0993 to 0.503]

10. Primary Outcome: Frequency of CD4+Foxp3- Expressing CD45RA and/or CTLA4 and/or OX40
Description: The frequency was assessed based on the following range of markers: CD4, CD45RA, CTLA4, OX40 and anti-Foxp3.
Time Frame: At the time of the visit for each subject (i.e., Day 0)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Treg cells/million cells
Arm/Group | Immune Tolerant Patients Group | HBeAg Positive Group | Inactive Carriers Group | HBeAg Negative Group
Number analyzed (Participants) | 4 | 11 | 56 | 18
Treg cells/million cells
  CD4+FOXP3- | 94.45 [91.9 to 98.2] | 93.9 [93.3 to 94.8] | 95.395 [93.85 to 96.645] | 94.95 [94 to 96.8]
  CD4+FOXP3-CD45RA+ | 45.2 [19.455 to 52.1] | 46.4 [37.1 to 53] | 36.05 [24.055 to 46.25] | 31.55 [22.2 to 38.9]
  CD4+FOXP3-CD45RA+CTLA4+OX40- | 0.2755 [0.0746 to 0.411] | 0.263 [0.212 to 0.456] | 0.2505 [0.0902 to 0.4915] | 0.265 [0.0806 to 0.475]
  CD4+FOXP3-CD45RA+CTLA4-OX40+ | 0.1715 [0.0816 to 0.1975] | 0.287 [0.128 to 0.488] | 0.1645 [0.0503 to 0.5495] | 0.243 [0.11 to 0.519]
  CD4+FOXP3-CD45RA+CTLA4-OX40- | 44.55 [18.9001 to 51.55] | 46 [36.7 to 52] | 34.4 [23.4 to 44.55] | 25.5 [18 to 35.4]
  CD4+FOXP3-CD45RA-CTLA4+OX40+ | 0.508 [0.2425 to 50.0535] | 0.242 [0.167 to 0.434] | 0.2645 [0.0736 to 0.619] | 0.6175 [0.31 to 1.37]
  CD4+FOXP3-CD45RA-CTLA4+OX40- | 2.35 [0.9599 to 2.865] | 1.87 [1.52 to 2.54] | 2.39 [1.79 to 3.34] | 1.845 [1.36 to 3.58]
  CD4+FOXP3-CD45RA-CTLA4-OX40+ | 3.035 [1.2051 to 4.495] | 2.48 [0.763 to 4.36] | 1.78 [0.603 to 5.855] | 4.015 [1.71 to 11.3]
  CD4+FOXP3-CD45RA-CTLA4-OX40- | 41.25 [19.5529 to 49.1] | 51.4 [39.7 to 58.4] | 53.05 [47 to 66.8] | 56.05 [51.4 to 68.2]
  CD4+FOXP3-CTLA4+ | 3.825 [2.92 to 52.015] | 2.34 [2.13 to 3.62] | 3.4 [2.14 to 4.52] | 3.55 [2 to 6.47]
  CD4+FOXP3-OX40+ | 5.235 [3.5 to 53.095] | 3.23 [1.34 to 5.2] | 2.27 [0.858 to 7.995] | 5.675 [2.65 to 13.1]
  CD4+polypositives FOXP3-CD45RA+CTLA4+OX40 | 0.0488 [0.0392 to 0.2813] | 0.0366 [0.0252 to 0.0662] | 0.0359 [0.0195 to 0.0803] | 0.0646 [0.0349 to 0.126]

11. Primary Outcome: Frequency of HBs- and HBc-specific CD4+Foxp3+ Expressing CD69 and/or LAP in Fresh Samples
Description: The frequency was assessed based on the following range of markers: CD4, CD69, LAP and anti-Foxp3.
Time Frame: At the time of the visit for each subject (i.e., Day 0)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Treg cells/million cells
Arm/Group | Immune Tolerant Patients Group | HBeAg Positive Group | Inactive Carriers Group | HBeAg Negative Group
Number analyzed (Participants) | 4 | 9 | 47 | 18
Treg cells/million cells
  HBc CD4+FOXP3+: number analyzed (Participants) | 3 | 9 | 47 | 18
  HBc CD4+FOXP3+ | 0.35 [0.26 to 0.36] | 0.21 [0.0001 to 0.53] | 0.42 [0.07 to 0.67] | 0.52 [0.12 to 0.81]
  HBc CD4+FOXP3+CD69+: number analyzed (Participants) | 3 | 9 | 47 | 18
  HBc CD4+FOXP3+CD69+ | 0.0001 [0.0001 to 0.0001] | 0.51 [0.08 to 1.08] | 0.84 [0.0001 to 2.8] | 1.0115 [0.0001 to 1.56]
  HBc CD4+FOXP3+LAP+: number analyzed (Participants) | 3 | 9 | 47 | 18
  HBc CD4+FOXP3+LAP+ | 0.0001 [0.0001 to 0.08] | 0.02 [0.0001 to 0.087] | 0.04 [0.0001 to 0.296] | 0.0001 [0.0001 to 0.158]
  HBc CD4+FOXP3+CD69+LAP+: number analyzed (Participants) | 3 | 9 | 47 | 18
  HBc CD4+FOXP3+CD69+LAP+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.072] | 0.082 [0.0001 to 0.32] | 0.0001 [0.0001 to 0.128]
  HBc CD4+FOXP3+CD69+LAP-: number analyzed (Participants) | 3 | 9 | 47 | 18
  HBc CD4+FOXP3+CD69+LAP- | 0.0001 [0.0001 to 0.55] | 0.69 [0.21 to 1.14] | 1.09 [0.0001 to 2.54] | 0.9815 [0.0001 to 1.93]
  HBc CD4+FOXP3+CD69-LAP+: number analyzed (Participants) | 3 | 9 | 47 | 18
  HBc CD4+FOXP3+CD69-LAP+ | 0.049 [0.0001 to 0.597] | 0.002 [0.0001 to 0.091] | 0.013 [0.0001 to 0.149] | 0.0086 [0.0001 to 0.194]
  HBc CD4+FOXP3+CD69-LAP-: number analyzed (Participants) | 3 | 9 | 47 | 18
  HBc CD4+FOXP3+CD69-LAP- | 0.6 [0.3 to 1.3] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.1] | 0.0001 [0.0001 to 0.1]
  HBs CD4+FOXP3+: number analyzed (Participants) | 4 | 9 | 44 | 18
  HBs CD4+FOXP3+ | 0.305 [0.0801 to 0.675] | 0.25 [0.0001 to 0.55] | 0.0101 [0.0001 to 0.2] | 0.16 [0.0001 to 0.66]
  HBs CD4+FOXP3+CD69+: number analyzed (Participants) | 4 | 9 | 44 | 18
  HBs CD4+FOXP3+CD69+ | 2.0101 [0.0001 to 4.135] | 0.95 [0.02 to 1.29] | 0.905 [0.0451 to 1.885] | 0.5315 [0.0001 to 2.45]
  HBs CD4+FOXP3+LAP+: number analyzed (Participants) | 4 | 9 | 44 | 18
  HBs CD4+FOXP3+LAP+ | 1.184 [0.5501 to 1.984] | 0.07 [0.0001 to 0.641] | 0.107 [0.0001 to 0.5965] | 0.0476 [0.0001 to 0.489]
  HBs CD4+FOXP3+CD69+LAP+: number analyzed (Participants) | 4 | 9 | 44 | 18
  HBs CD4+FOXP3+CD69+LAP+ | 0.2201 [0.0001 to 1.395] | 0.0001 [0.0001 to 0.299] | 0.0001 [0.0001 to 0.149] | 0.0001 [0.0001 to 0.23]
  HBs CD4+FOXP3+CD69+LAP-: number analyzed (Participants) | 4 | 9 | 44 | 18
  HBs CD4+FOXP3+CD69+LAP- | 1.025 [0.0751 to 3.055] | 0.65 [0.34 to 1.31] | 1.01 [0.4535 to 2.2] | 0.5215 [0.0001 to 2.16]
  HBs CD4+FOXP3+CD69-LAP+: number analyzed (Participants) | 4 | 9 | 44 | 18
  HBs CD4+FOXP3+CD69-LAP+ | 0.5065 [0.1731 to 1.064] | 0.033 [0.0001 to 0.346] | 0.0805 [0.0001 to 0.392] | 0.1335 [0.0001 to 0.394]
  HBs CD4+FOXP3+CD69-LAP-: number analyzed (Participants) | 4 | 9 | 44 | 18
  HBs CD4+FOXP3+CD69-LAP- | 0.0001 [0.0001 to 0.4501] | 0.0001 [0.0001 to 0.1] | 0.0001 [0.0001 to 0.0501] | 0.0001 [0.0001 to 0.6]

12. Primary Outcome: Frequency of HBs- and HBc-specific CD4+Foxp3- Expressing CD69 and/or LAP in Fresh Samples
Description: The frequency was assessed based on the following range of markers: CD4, CD69, LAP and anti-Foxp3.
Time Frame: At the time of the visit for each subject (i.e., Day 0)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Treg cells/million cells
Arm/Group | Immune Tolerant Patients Group | HBeAg Positive Group | Inactive Carriers Group | HBeAg Negative Group
Number analyzed (Participants) | 4 | 11 | 56 | 19
Treg cells/million cells
  HBc CD4+FOXP3- | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.5] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD4+FOXP3-CD69+ | 0.0001 [0.0001 to 0.6246] | 0.16 [0.0001 to 0.22] | 0.28 [0.0001 to 1.26] | 0.25 [0.053 to 0.91]
  HBc CD4+FOXP3-LAP+ | 0.0051 [0.0001 to 0.05] | 0.02 [0.0001 to 0.08] | 0.0345 [0.0001 to 0.147] | 0.0001 [0.0001 to 0.104]
  HBc CD4+FOXP3-CD69+LAP+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.037] | 0.01 [0.0001 to 0.0515] | 0.0126 [0.0001 to 0.0373]
  HBc CD4+FOXP3-CD69+LAP- | 0.33 [0.1351 to 0.828] | 0.15 [0.0001 to 0.27] | 0.185 [0.0001 to 1.245] | 0.279 [0.078 to 0.94]
  HBc CD4+FOXP3-CD69-LAP+ | 0.0672 [0.0158 to 0.1165] | 0.025 [0.0001 to 0.0675] | 0.0165 [0.0001 to 0.108] | 0.0001 [0.0001 to 0.0642]
  HBc CD4+FOXP3-CD69-LAP- | 0.2501 [0.0001 to 1.25] | 0.0001 [0.0001 to 0.2] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.1]
  HBs CD4+FOXP3- | 0.0001 [0.0001 to 0.0501] | 0.1 [0.0001 to 0.5] | 0.0001 [0.0001 to 0.35] | 0.0001 [0.0001 to 0.0001]
  HBs CD4+FOXP3-CD69+ | 0.0001 [0.0001 to 1.4146] | 0.0001 [0.0001 to 0.0001] | 0.068 [0.0001 to 0.475] | 0.07 [0.0001 to 0.24]
  HBs CD4+FOXP3-LAP+ | 0.2251 [0.0001 to 0.555] | 0.0913 [0.0001 to 0.219] | 0.0993 [0.0001 to 0.3005] | 0.0001 [0.0001 to 0.328]
  HBs CD4+FOXP3-CD69+LAP+ | 0.0001 [0.0001 to 0.0309] | 0.0001 [0.0001 to 0.044] | 0.0001 [0.0001 to 0.0229] | 0.0057 [0.0001 to 0.075]
  HBs CD4+FOXP3-CD69+LAP- | 0.1901 [0.0001 to 1.573] | 0.0001 [0.0001 to 0.011] | 0.1 [0.0001 to 0.4465] | 0.087 [0.0001 to 0.233]
  HBs CD4+FOXP3-CD69-LAP+ | 0.334 [0.0736 to 0.5597] | 0.173 [0.0001 to 0.208] | 0.1011 [0.0001 to 0.2795] | 0.046 [0.0001 to 0.244]
  HBs CD4+FOXP3-CD69-LAP- | 0.45 [0.0501 to 1] | 0.1 [0.0001 to 0.5] | 0.0001 [0.0001 to 0.1] | 0.0001 [0.0001 to 0.0001]

13. Primary Outcome: Frequency of HBc-specific CD4+Foxp3+ Expressing CD69 and/or LAP in Frozen Samples
Description: The frequency was assessed based on the following range of markers: CD4, CD69, LAP and anti-Foxp3.
Time Frame: At the time of the visit for each subject (i.e., Day 0)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Treg cells/million cells
Arm/Group | Immune Tolerant Patients Group | HBeAg Positive Group | Inactive Carriers Group | HBeAg Negative Group
Number analyzed (Participants) | 1 | 4 | 26 | 9
Treg cells/million cells
  CD4+FOXP3+CD69+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.2301] | 0.0001 [0.0001 to 0.62] | 0.8 [0.0001 to 2.2]
  CD4+FOXP3+LAP+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.1671] | 0.0001 [0.0001 to 0.067] | 0.29 [0.0001 to 0.67]
  CD4+FOXP3+CD69+LAP+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.1915] | 0.0001 [0.0001 to 0.014] | 0.259 [0.01 to 0.61]
  CD4+FOXP3+CD69+LAP- | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0351] | 0.0001 [0.0001 to 0.67] | 0.2 [0.0001 to 2.2]
  CD4+FOXP3+CD69-LAP+ | 0.74 [0.74 to 0.74] | 0.0001 [0.0001 to 0.0001] | 0.055 [0.0001 to 0.25] | 0.06 [0.0001 to 0.274]

14. Secondary Outcome: Frequency of CD4+ Expressing CD40-L and/or Interferon-gamma (IFNg) and/or Interleukin 2 (IL-2) and/or IL-17 in Fresh Samples
Description: The frequency was assessed based on the following range of markers: CD4, CD40-L, IFNg, IL-2 and IL-17.
  Note: The precision of the measure (i.e., four decimals) of median and inter-quartile range is not sufficient to distinguish between the values median, lower and upper limits of inter-quartile range for some of the data presented within the table below (e.g., median=0.0001 and inter-quartile range=0.0001 to 0.0001).
Time Frame: At the time of the visit for each subject (i.e., Day 0)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Treg cells/million cells
Arm/Group | Immune Tolerant Patients Group | HBeAg Positive Group | Inactive Carriers Group | HBeAg Negative Group
Number analyzed (Participants) | 4 | 11 | 57 | 20
Treg cells/million cells
  HBc CD4+CD40L+ | 0.0181 [0.0056 to 0.0294] | 0.0032 [0.0001 to 0.0209] | 0.0013 [0.0001 to 0.0255] | 0.0135 [0.0001 to 0.0271]
  HBc CD4+IFNg+ | 0.0164 [0.0001 to 0.038] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD4+IL2+ | 0.0044 [0.0001 to 0.0255] | 0.0001 [0.0001 to 0.0023] | 0.0014 [0.0001 to 0.012] | 0.0004 [0.0001 to 0.0066]
  HBc CD4+IL17+ | 0.0128 [0.0015 to 0.0277] | 0.0025 [0.0001 to 0.009] | 0.0004 [0.0001 to 0.0043] | 0.0014 [0.0001 to 0.0089]
  HBc CD4+CD40L+IL2+IFNg+IL17+ | 0.0001 [0.0001 to 0.0017] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD4+CD40L+IL2+IFNg+IL17- | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD4+CD40L+IL2-IFNg+IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD4+CD40L+IL2-IFNg+IL17- | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD4+CD40L+IL2+IFNg-IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD4+CD40L+IL2+IFNg-IL17- | 0.0018 [0.0007 to 0.003] | 0.0001 [0.0001 to 0.0018] | 0.0025 [0.0001 to 0.0066] | 0.0011 [0.0001 to 0.0036]
  HBc CD4+CD40L+IL2-IFNg-IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0024] | 0.0001 [0.0001 to 0.002] | 0.0001 [0.0001 to 0.0001]
  HBc CD4+CD40L+IL2-IFNg-IL17- | 0.0158 [0.0051 to 0.026] | 0.0023 [0.0001 to 0.0122] | 0.0013 [0.0001 to 0.0216] | 0.0113 [0.0001 to 0.0259]
  HBc CD4+CD40L-IL2+IFNg+IL17+ | 0.0038 [0.0001 to 0.024] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD4+CD40L-IL2+IFNg+IL17- | 0.0001 [0.0001 to 0.0017] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD4+CD40L-IL2-IFNg+IL17+ | 0.0001 [0.0001 to 0.0088] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD4+CD40L-IL2-IFNg+IL17- | 0.0023 [0.0001 to 0.0072] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0006]
  HBc CD4+CD40L-IL2+IFNg-IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0012] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0002]
  HBc CD4+CD40L-IL2+IFNg-IL17- | 0.0001 [0.0001 to 0.0013] | 0.0001 [0.0001 to 0.0002] | 0.0001 [0.0001 to 0.002] | 0.0001 [0.0001 to 0.0023]
  HBc CD4+CD40L-IL2-IFNg-IL17+ | 0.0006 [0.0001 to 0.0015] | 0.0001 [0.0001 to 0.0018] | 0.0012 [0.0001 to 0.0054] | 0.0022 [0.0001 to 0.0036]
  HBs CD4+CD40L+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD4+CD40L+ | 0.0001 [0.0001 to 0.0051] | 0.0001 [0.0001 to 0.0062] | 0.0001 [0.0001 to 0.0127] | 0.0053 [0.0001 to 0.0207]
  HBs CD4+IFNg+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD4+IFNg+ | 0.0011 [0.0001 to 0.0143] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBs CD4+IL2+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD4+IL2+ | 0.0049 [0.0001 to 0.011] | 0.0064 [0.0001 to 0.0191] | 0.0021 [0.0001 to 0.0151] | 0.0001 [0.0001 to 0.0062]
  HBs CD4+IL17+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD4+IL17+ | 0.0013 [0.0001 to 0.0165] | 0.0058 [0.0001 to 0.0486] | 0.0001 [0.0001 to 0.0024] | 0.0002 [0.0001 to 0.0061]
  HBs CD4+CD40L+IL2+IFNg+IL17+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD4+CD40L+IL2+IFNg+IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBs CD4+CD40L+IL2+IFNg+IL17-: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD4+CD40L+IL2+IFNg+IL17- | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBs CD4+CD40L+IL2-IFNg+IL17+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD4+CD40L+IL2-IFNg+IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBs CD4+CD40L+IL2-IFNg+IL17-: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD4+CD40L+IL2-IFNg+IL17- | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBs CD4+CD40L+IL2+IFNg-IL17+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD4+CD40L+IL2+IFNg-IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0013] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBs CD4+CD40L+IL2+IFNg-IL17-: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD4+CD40L+IL2+IFNg-IL17- | 0.0001 [0.0001 to 0.0007] | 0.0015 [0.0001 to 0.0038] | 0.0001 [0.0001 to 0.0028] | 0.0001 [0.0001 to 0.0021]
  HBs CD4+CD40L+IL2-IFNg-IL17+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD4+CD40L+IL2-IFNg-IL17+ | 0.0001 [0.0001 to 0.0007] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBs CD4+CD40L+IL2-IFNg-IL17-: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD4+CD40L+IL2-IFNg-IL17- | 0.0001 [0.0001 to 0.0051] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0095] | 0.0041 [0.0001 to 0.0181]
  HBs CD4+CD40L-IL2+IFNg+IL17+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD4+CD40L-IL2+IFNg+IL17+ | 0.0025 [0.0001 to 0.0075] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBs CD4+CD40L-IL2+IFNg+IL17-: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD4+CD40L-IL2+IFNg+IL17- | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBs CD4+CD40L-IL2-IFNg+IL17+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD4+CD40L-IL2-IFNg+IL17+ | 0.0001 [0.0001 to 0.0068] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBs CD4+CD40L-IL2-IFNg+IL17-: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD4+CD40L-IL2-IFNg+IL17- | 0.0001 [0.0001 to 0.0015] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBs CD4+CD40L-IL2+IFNg-IL17+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD4+CD40L-IL2+IFNg-IL17+ | 0.0001 [0.0001 to 0.0036] | 0.0001 [0.0001 to 0.004] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBs CD4+CD40L-IL2+IFNg-IL17-: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD4+CD40L-IL2+IFNg-IL17- | 0.0001 [0.0001 to 0.0044] | 0.0001 [0.0001 to 0.0143] | 0.0017 [0.0001 to 0.0108] | 0.0001 [0.0001 to 0.0035]
  HBs CD4+CD40L-IL2-IFNg-IL17+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD4+CD40L-IL2-IFNg-IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0019 [0.0001 to 0.004] | 0.0001 [0.0001 to 0.0021] | 0.0001 [0.0001 to 0.001]

15. Secondary Outcome: Frequency of Cluster of Differentiation 8 (CD8+) Expressing CD40-L and/or IFNg and/or IL-2 and/or IL-17 in Fresh Samples
Description: The frequency was assessed based on the following range of markers: CD8, CD40-L, IFNg, IL-2 and IL-17.
  Note: The precision of the measure (i.e., four decimals) of median and inter-quartile range is not sufficient to distinguish between the values median, lower and upper limits of inter-quartile range for some of the data presented within the table below (e.g., median=0.0001 and inter-quartile range=0.0001 to 0.0001).
Time Frame: At the time of the visit for each subject (i.e., Day 0)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Treg cells/million cells
Arm/Group | Immune Tolerant Patients Group | HBeAg Positive Group | Inactive Carriers Group | HBeAg Negative Group
Number analyzed (Participants) | 4 | 11 | 57 | 20
Treg cells/million cells
  HBc CD8+CD40L+ | 0.004 [0.002 to 0.0071] | 0.0034 [0.0001 to 0.0106] | 0.0002 [0.0001 to 0.0128] | 0.0065 [0.0001 to 0.0098]
  HBc CD8+IFNg+ | 0.0346 [0.0197 to 0.0609] | 0.003 [0.0001 to 0.0117] | 0.0001 [0.0001 to 0.0048] | 0.0003 [0.0001 to 0.0197]
  HBc CD8+IL2+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0053] | 0.0001 [0.0001 to 0.0052] | 0.001 [0.0001 to 0.0101]
  HBc CD8+IL17+ | 0.0001 [0.0001 to 0.0153] | 0.0001 [0.0001 to 0.0345] | 0.0021 [0.0001 to 0.0523] | 0.0001 [0.0001 to 0.0097]
  HBc CD8+CD40L+IL2+IFNg+IL17+ | 0.0001 [0.0001 to 0.0005] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD8+CD40L+IL2+IFNg+IL17- | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD8+CD40L+IL2-IFNg+IL17+ | 0.0001 [0.0001 to 0.0016] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD8+CD40L+IL2-IFNg+IL17- | 0.0001 [0.0001 to 0.0017] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD8+CD40L+IL2+IFNg-IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD8+CD40L+IL2+IFNg-IL17- | 0.0001 [0.0001 to 0.0016] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD8+CD40L+IL2-IFNg-IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD8+CD40L+IL2-IFNg-IL17- | 0.0039 [0.002 to 0.007] | 0.0052 [0.0001 to 0.0106] | 0.0002 [0.0001 to 0.0126] | 0.0066 [0.0001 to 0.0111]
  HBc CD8+CD40L-IL2+IFNg+IL17+ | 0.0001 [0.0001 to 0.0005] | 0.0001 [0.0001 to 0.0034] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD8+CD40L-IL2+IFNg+IL17- | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0014]
  HBc CD8+CD40L-IL2-IFNg+IL17+ | 0.0034 [0.0001 to 0.0155] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD8+CD40L-IL2-IFNg+IL17- | 0.0251 [0.0115 to 0.0548] | 0.0001 [0.0001 to 0.0097] | 0.0001 [0.0001 to 0.0048] | 0.0008 [0.0001 to 0.0113]
  HBc CD8+CD40L-IL2+IFNg-IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.001]
  HBc CD8+CD40L-IL2+IFNg-IL17- | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0035] | 0.0001 [0.0001 to 0.0041]
  HBc CD8+CD40L-IL2-IFNg-IL17+ | 0.0001 [0.0001 to 0.0025] | 0.0001 [0.0001 to 0.004] | 0.0021 [0.0001 to 0.045] | 0.0001 [0.0001 to 0.0044]
  HBs CD8+CD40L+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD8+CD40L+ | 0.0046 [0.0005 to 0.009] | 0.0001 [0.0001 to 0.0057] | 0.0001 [0.0001 to 0.0118] | 0.0002 [0.0001 to 0.0073]
  HBs CD8+IFNg+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD8+IFNg+ | 0.0167 [0.0087 to 0.0324] | 0.0001 [0.0001 to 0.0064] | 0.0027 [0.0001 to 0.0155] | 0.0001 [0.0001 to 0.0117]
  HBs CD8+IL2+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD8+IL2+ | 0.0001 [0.0001 to 0.011] | 0.0001 [0.0001 to 0.031] | 0.0013 [0.0001 to 0.0066] | 0.0001 [0.0001 to 0.0049]
  HBs CD8+IL17+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD8+IL17+ | 0.0001 [0.0001 to 0.0158] | 0.0001 [0.0001 to 0.0448] | 0.0015 [0.0001 to 0.0462] | 0.0001 [0.0001 to 0.0395]
  HBs CD8+CD40L+IL2+IFNg+IL17+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD8+CD40L+IL2+IFNg+IL17+ | 0.0001 [0.0001 to 0.0026] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBs CD8+CD40L+IL2+IFNg+IL17-: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD8+CD40L+IL2+IFNg+IL17- | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBs CD8+CD40L+IL2-IFNg+IL17+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD8+CD40L+IL2-IFNg+IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBs CD8+CD40L+IL2-IFNg+IL17-: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD8+CD40L+IL2-IFNg+IL17- | 0.0001 [0.0001 to 0.0019] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBs CD8+CD40L+IL2+IFNg-IL17+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD8+CD40L+IL2+IFNg-IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBs CD8+CD40L+IL2+IFNg-IL17-: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD8+CD40L+IL2+IFNg-IL17- | 0.0017 [0.0001 to 0.0074] | 0.0001 [0.0001 to 0.0003] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBs CD8+CD40L+IL2-IFNg-IL17+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD8+CD40L+IL2-IFNg-IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBs CD8+CD40L+IL2-IFNg-IL17-: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD8+CD40L+IL2-IFNg-IL17- | 0.0046 [0.0005 to 0.0083] | 0.0001 [0.0001 to 0.0083] | 0.0001 [0.0001 to 0.0106] | 0.0002 [0.0001 to 0.0038]
  HBs CD8+CD40L-IL2+IFNg+IL17+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD8+CD40L-IL2+IFNg+IL17+ | 0.0001 [0.0001 to 0.0139] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBs CD8+CD40L-IL2+IFNg+IL17-: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD8+CD40L-IL2+IFNg+IL17- | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBs CD8+CD40L-IL2-IFNg+IL17+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD8+CD40L-IL2-IFNg+IL17+ | 0.0016 [0.0001 to 0.0035] | 0.0001 [0.0001 to 0.0038] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBs CD8+CD40L-IL2-IFNg+IL17-: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD8+CD40L-IL2-IFNg+IL17- | 0.0126 [0.0056 to 0.0198] | 0.0001 [0.0001 to 0.0067] | 0.0001 [0.0001 to 0.0126] | 0.0001 [0.0001 to 0.0348]
  HBs CD8+CD40L-IL2+IFNg-IL17+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD8+CD40L-IL2+IFNg-IL17+ | 0.0001 [0.0001 to 0.0019] | 0.0001 [0.0001 to 0.0019] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0009]
  HBs CD8+CD40L-IL2+IFNg-IL17-: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD8+CD40L-IL2+IFNg-IL17- | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0041] | 0.0001 [0.0001 to 0.0066] | 0.0001 [0.0001 to 0.0001]
  HBs CD8+CD40L-IL2-IFNg-IL17+: number analyzed (Participants) | 4 | 11 | 56 | 20
  HBs CD8+CD40L-IL2-IFNg-IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.029] | 0.0026 [0.0001 to 0.0446] | 0.0001 [0.0001 to 0.0269]

16. Secondary Outcome: Frequency of CD4+ Expressing CD40-L and/or IFNg and/or IL-2 and/or IL-17 in Frozen Samples
Description: as for outcome 14
Time Frame: At the time of the visit for each subject (i.e., Day 0)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Treg cells/million cells
Arm/Group | Immune Tolerant Patients Group | HBeAg Positive Group | Inactive Carriers Group | HBeAg Negative Group
Number analyzed (Participants) | 2 | 7 | 40 | 11
Treg cells/million cells
  HBc CD4+CD40L+ | 0.0048 [0.0001 to 0.0095] | 0.108 [0.0148 to 0.337] | 0.0336 [0.0001 to 0.2448] | 0.032 [0.0001 to 0.453]
  HBc CD4+IFNg+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0099] | 0.0001 [0.0001 to 0.0097] | 0.0001 [0.0001 to 0.0001]
  HBc CD4+IL2+ | 0.0161 [0.0001 to 0.0321] | 0.0128 [0.0001 to 0.0486] | 0.0033 [0.0001 to 0.0245] | 0.0083 [0.0001 to 0.0368]
  HBc CD4+IL17+ | 0.0063 [0.0001 to 0.0124] | 0.0012 [0.0001 to 0.0046] | 0.0047 [0.0002 to 0.0154] | 0.0037 [0.0007 to 0.0139]
  HBc CD4+CD40L+IL2+IFNg+IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD4+CD40L+IL2+IFNg+IL17- | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD4+CD40L+IL2-IFNg+IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD4+CD40L+IL2-IFNg+IL17- | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0014] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0007]
  HBc CD4+CD40L+IL2+IFNg-IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD4+CD40L+IL2+IFNg-IL17- | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0009] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD4+CD40L+IL2-IFNg-IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD4+CD40L+IL2-IFNg-IL17- | 0.0048 [0.0001 to 0.0095] | 0.105 [0.0148 to 0.347] | 0.031 [0.0001 to 0.2438] | 0.031 [0.0001 to 0.45]
  HBc CD4+CD40L-IL2+IFNg+IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD4+CD40L-IL2+IFNg+IL17- | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0008] | 0.0001 [0.0001 to 0.0001]
  HBc CD4+CD40L-IL2-IFNg+IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD4+CD40L-IL2-IFNg+IL17- | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0085] | 0.0001 [0.0001 to 0.0095] | 0.0001 [0.0001 to 0.0001]
  HBc CD4+CD40L-IL2+IFNg-IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD4+CD40L-IL2+IFNg-IL17- | 0.0161 [0.0001 to 0.0321] | 0.0104 [0.0001 to 0.0522] | 0.0022 [0.0001 to 0.0213] | 0.0083 [0.0001 to 0.0348]
  HBc CD4+CD40L-IL2-IFNg-IL17+ | 0.0063 [0.0001 to 0.0124] | 0.0012 [0.0001 to 0.0057] | 0.0048 [0.0001 to 0.0158] | 0.0039 [0.0007 to 0.0139]

17. Secondary Outcome: Frequency of CD8+ Expressing CD40-L and/or IFNg and/or IL-2 and/or IL-17 in Frozen Samples
Description: The frequency was assessed based on the following range of markers: CD8, CD40L, IFNg, IL-2 and IL-17.
  Note: The precision of the measure (i.e., four decimals) of median and inter-quartile range is not sufficient to distinguish between the values median, lower and upper limits of inter-quartile range for some of the data presented within the table below (e.g., median=0.0001 and inter-quartile range=0.0001 to 0.0001).
Time Frame: At the time of the visit for each subject (i.e., Day 0)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Treg cells/million cells
Arm/Group | Immune Tolerant Patients Group | HBeAg Positive Group | Inactive Carriers Group | HBeAg Negative Group
Number analyzed (Participants) | 2 | 7 | 40 | 11
Treg cells/million cells
  HBc CD8+CD40L+ | 0.0001 [0.0001 to 0.0001] | 0.0556 [0.0001 to 0.1472] | 0.0001 [0.0001 to 0.0265] | 0.0035 [0.0001 to 0.0193]
  HBc CD8+IFNg+ | 0.0246 [0.0127 to 0.0365] | 0.0001 [0.0001 to 0.0239] | 0.0001 [0.0001 to 0.0248] | 0.0002 [0.0001 to 0.023]
  HBc CD8+IL2+ | 0.0448 [0.0078 to 0.0819] | 0.0001 [0.0001 to 0.0195] | 0.0004 [0.0001 to 0.015] | 0.0042 [0.0001 to 0.0105]
  HBc CD8+IL17+ | 0.1191 [0.0001 to 0.238] | 0.0001 [0.0001 to 0.0768] | 0.0058 [0.0001 to 0.0716] | 0.0075 [0.0001 to 0.15]
  HBc CD8+CD40L+IL2+IFNg+IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD8+CD40L+IL2+IFNg+IL17- | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD8+CD40L+IL2-IFNg+IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD8+CD40L+IL2-IFNg+IL17- | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD8+CD40L+IL2+IFNg-IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD8+CD40L+IL2+IFNg-IL17- | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD8+CD40L+IL2-IFNg-IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD8+CD40L+IL2-IFNg-IL17- | 0.0001 [0.0001 to 0.0001] | 0.0556 [0.0001 to 0.1554] | 0.0001 [0.0001 to 0.0277] | 0.0035 [0.0001 to 0.0193]
  HBc CD8+CD40L-IL2+IFNg+IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD8+CD40L-IL2+IFNg+IL17- | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0011] | 0.0001 [0.0001 to 0.0012]
  HBc CD8+CD40L-IL2-IFNg+IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD8+CD40L-IL2-IFNg+IL17- | 0.0246 [0.0127 to 0.0365] | 0.0001 [0.0001 to 0.0227] | 0.0001 [0.0001 to 0.0217] | 0.0001 [0.0001 to 0.023]
  HBc CD8+CD40L-IL2+IFNg-IL17+ | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001] | 0.0001 [0.0001 to 0.0001]
  HBc CD8+CD40L-IL2+IFNg-IL17- | 0.0448 [0.0078 to 0.0819] | 0.0001 [0.0001 to 0.0109] | 0.0053 [0.0001 to 0.0153] | 0.0002 [0.0001 to 0.0088]
  HBc CD8+CD40L-IL2-IFNg-IL17+ | 0.1166 [0.0001 to 0.233] | 0.0001 [0.0001 to 0.0768] | 0.0058 [0.0001 to 0.0761] | 0.0075 [0.0001 to 0.152]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) related to study participation or to GSK concomitant products were collected during the study: from the time each subject consented to participate in the study up to study conclusion (i.e. during an approximate period of 22 months).
Description: Other (non-serious) Adverse Events were not collected in the study.
Arm/Group | Immune Tolerant Patients Group | HBeAg Positive Group | Inactive Carriers Group | HBeAg Negative Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/11 | 0/60 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/11 | 0/60 | 0/21
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.